CLINICAL TRIAL: NCT01096485
Title: Open-label, Randomized, Crossover Study to Compare the Bioavailability of One Coated Tablet of Opxion® (Levonorgestrel 1.5 mg From Bayer de Mexico) vs. Two Tablets of Postday® (Levonorgestrel 0.75 mg From Investigacion Farmaceutica), in Healthy Volunteers
Brief Title: Cross-over Study to Prove Bioequivalence Between Two Oral Formulations of Levonorgestrel
Acronym: LEVEQ-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer de Mexico S.A. de C.V.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 13956
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Contraception; Contraception, Postcoital
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levonorgestrel Emergency Pill (BAY86-5028/Opxion)
- Arm 2 (Active Comparator)
  Interventions: Drug: Levonorgestrel (Postday)

INTERVENTIONS:
Drug: Levonorgestrel Emergency Pill (BAY86-5028/Opxion) — Single dose of 1.5 mg coated tablet
  Arms: Arm 1
Drug: Levonorgestrel (Postday) — Single dose of two 0.75 mg tablets
  Arms: Arm 2

SUMMARY:
A single dose, two treatments (Postday and Opxion), two periods, two sequences, crossover, randomized, prospective design was chosen with a washout of 21 days between the two study periods. Treatment groups were balanced with the same number of male healthy volunteers who were randomly assigned to the study drug administration sequences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers age between 18 and 55 years old with normal vital signs, electrocardiogram (ECG), blood chemistry, liver function profile and urinalysis.

Exclusion Criteria:

* History of illnesses or any organic abnormalities that could affect the results of the study.
* History of abuse tobacco or alcohol or regular use of recreational or therapeutic drugs.
* Subjects that have taken any medication within 14 days or that are in an elimination period of less than 7 half-lives (whichever is longest) before study startup.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Least square estimator of average maximum plasmatic concentration (log transformed) | After 2 months
Least square estimator of area under the pharmacokinetic curve (log transformed) | After 2 months

SECONDARY OUTCOMES:
Time at which maximum concentration is reached | After 2 months
Area under the pharmacokinetic curve from time=0 to time of last blood sample | After 2 months
Clearance constant of plasmatic concentration of study drug | After 2 months
Half life of plasmatic concentration of study drug | After 2 months
Adverse events collection | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Morelia, Michoacán, Mexico